CLINICAL TRIAL: NCT02999659
Title: Impact of Acute Cerebral Diseases on the Autonomous Nervous System: Progression and Correlation to Therapy and Outcome
Acronym: Pupillometry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Gerrit Alexander Schubert, apl. Prof. Dr. med. Gerrit Alexander Schubert, RWTH Aachen University
Other Study IDs: 16-035
Record Dates: First submitted 2016-12-19; First posted 2016-12-21 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Pupillary Function, Abnormal; Cerebral Aneurysm
Keywords: pupillometry; autonomous nerve system
MeSH Terms: conditions — Pupil Disorders; Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group: The control group implies patients with non-acute cerebral disease (e.g. cerebral aneurysm without symptoms). The pupilometer data are once collected during ambulant routine examination. The patients do not undergo any further study related examinations.
  Interventions: Device: Pupilometer
- Treatment group: The treatment group implies patients with an acute cerebral disease ensured by CT, MRI or spinal tap. Pupillometry measurements are done during neurological routine examinations. Generally, during the initial diagnosis examination, followed by daily routine measurements and after 3 and 6 month upon hospital discharge.
  Interventions: Device: Pupilometer

INTERVENTIONS:
Device: Pupilometer — Device to measure change in pupil diameter due to a defined light stimulus.

SUMMARY:
The pupilometer determines the alteration of the pupil diameter after a defined light stimulus. In this study data is collected from pupilometer measurements of patients with an acute cerebral disease. The measurements take place during daily neurological routine examinations. The values are compared to outcomes resulting from pupilometer measurements done on patients having not an acute cerebral disease (e.g. cerebral aneurysm without symptoms). The study aims to establish the not invasive method of pupillometry for detecting neurological degradations early.

DETAILED DESCRIPTION:
The pupilometer determines the alteration of the pupil diameter after a defined light stimulus providing information of the autonomic nerve system. The result collecting from pupillometry is objective and more precise than the subjective-visual evaluation of the pupil and its reactivity.

In this observational study data is collected from pupilometer measurements of patients with an acute cerebral disease. The measurements take place during neurological routine examinations. The first measurement is done during the initial diagnosing examination, followed by daily measurements and ending with measurements after 3 and 6 month upon hospital discharge. The values are compared to standard values resulting from pupilometer measurements done on patients having non-acute cerebral disease (e.g. cerebral aneurysm without symptoms). The study aims to establish the not invasive method of pupillometry for detecting neurological degradations early.

ELIGIBILITY:
Inclusion Criteria:

* male or female patient, age ≥ 18 years
* signed consent
* treatment group:
* patient with acute, cerebral disease verified by CT, MRI or spinal tap
* control group
* patient with non-acute cerebral disease like a new diagnosed aneurysm without symptoms

Exclusion Criteria:

* female or male patient aged < 18 years
* absent of signed consent
* persons who have a dependent or working relationship with the sponsor or investigator
* persons who are sheltered in an institution by juridical or governmental order
* concurrent participation in an other clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study includes male and female patients suffering from a acute (treatment group) or non-acute (control group) cerebral disease with a minimum age of 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-12; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Number of delayed cerebral ischemia (DCI) | 21 days
  DCI is defined as the development of new focal neurological signs and/or deterioration in level of consciousness, lasting for more than 1 h, or the appearance of new infarctions on CT or MRI.
Number of perfusion deficiency | 21 days

SECONDARY OUTCOMES:
Transcranial Doppler (TCD) -fluency increase [cm/s] | 21 days
  > 150 cm/s absolute or increase > 50 cm/s within 24 h
Digital subtraction angiography (DSA) | day 7 ± 2 d
  Detection of an angiographic vasospasm
Glasgow Outcome Score (GOS) | after 3 and 6 month
  Standardized and objective description of the degree of recovery of patients suffered from a cerebral disease.

CONTACTS AND LOCATIONS:
Overall Officials: Gerrit Alexander Schubert, Prof., Principal Investigator — Uniklinik RWTH Aachen
Locations (1):
- Uniklinik RWTH Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen JW, Gombart ZJ, Rogers S, Gardiner SK, Cecil S, Bullock RM. Pupillary reactivity as an early indicator of increased intracranial pressure: The introduction of the Neurological Pupil index. Surg Neurol Int. 2011;2:82. doi: 10.4103/2152-7806.82248. Epub 2011 Jun 21. PMID 21748035
- [Background] Ciurea AV, Palade C, Voinescu D, Nica DA. Subarachnoid hemorrhage and cerebral vasospasm - literature review. J Med Life. 2013 Jun 15;6(2):120-5. Epub 2013 Jun 25. PMID 23904869
- [Background] Cocker KD, Moseley MJ, Stirling HF, Fielder AR. Delayed visual maturation: pupillary responses implicate subcortical and cortical visual systems. Dev Med Child Neurol. 1998 Mar;40(3):160-2. doi: 10.1111/j.1469-8749.1998.tb15440.x. PMID 9566651
- [Background] Fountas KN, Kapsalaki EZ, Machinis TG, Boev AN, Robinson JS, Troup EC. Clinical implications of quantitative infrared pupillometry in neurosurgical patients. Neurocrit Care. 2006;5(1):55-60. doi: 10.1385/NCC:5:1:55. PMID 16960298
- [Background] Rowland MJ, Hadjipavlou G, Kelly M, Westbrook J, Pattinson KT. Delayed cerebral ischaemia after subarachnoid haemorrhage: looking beyond vasospasm. Br J Anaesth. 2012 Sep;109(3):315-29. doi: 10.1093/bja/aes264. PMID 22879655
- [Background] Toi H, Matsumoto N, Yokosuka K, Matsubara S, Hirano K, Uno M. Prediction of cerebral vasospasm using early stage transcranial Doppler. Neurol Med Chir (Tokyo). 2013;53(6):396-402. doi: 10.2176/nmc.53.396. PMID 23803618
- [Background] Larson MD, Singh V. Portable infrared pupillometry in critical care. Crit Care. 2016 Jun 22;20(1):161. doi: 10.1186/s13054-016-1349-7. PMID 27329287